CLINICAL TRIAL: NCT04912284
Title: Africa COVID-19 Vaccine Hesitancy: a Multi-country Cross-sectional Study
Brief Title: Africa COVID-19 Vaccine Hesitancy
Acronym: ACHES
Status: Completed | Type: Observational
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); University of Bamako (Other); Cheikh Anta Diop University, Senegal (Other); University of Sierra Leone (Other); Gamal Abdel Nasser University of Conakry (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-10550-BO-ff
Record Dates: First submitted 2021-05-31; First posted 2021-06-03 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Vaccine hesitancy; Vaccines; West Africa
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General population: Questionnaire administered to adult population
- Health care workers: Questionnaire administered to adult health care workers

SUMMARY:
Vaccine hesitancy is defined by the WHO's Strategic Advisory Group of Experts on Immunization as a 'delay in acceptance or refusal of vaccination despite availability of vaccination services'. This varies in form and intensity based on when and where it occurs and what vaccine is involved. Several prophylactic vaccines against COVID-19 are currently available. As the world is beginning the roll-out the first approved vaccines, little is known about people's potential acceptance of a COVID-19 vaccine in most of the African countries. ACHES (African COVID -19Vaccine Hesitancy) is an observational study aimed at measuring COVID-19 vaccine hesitancy in five west African countries and exploring causes behind the hesitancy with the main objective of informing guidelines for the proficient roll-out of the vaccines in the region.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) was declared a Public Health Emergency of International Concern by the World Health Organization (WHO) in March 2020. Although African countries seem to have weathered the pandemic relatively well so far, with fewer than one confirmed case for every thousand people and around 50,000 death, the African continent has now officially over two million- COVID-19- case threshold.

In 2015, WHO's Strategic Advisory Group of Experts on Immunization defined vaccine hesitancy as a 'delay in acceptance or refusal of vaccination despite availability of vaccination services', which can vary in form and intensity based on when and where it occurs and what vaccine is involved. Several prophylactic vaccines against COVID-19 are currently in development. As the world is beginning the roll-out the first approved vaccines, little is known about people's potential acceptance of a COVID-19 vaccine in most of the African countries. A recent study published in Nature provides results on the acceptability of vaccines in 19 of the 35 hardest hit countries worldwide. South Africa was the only African country included in the survey. An additional survey conducted in 15 African countries between August and December 2020, reveals that the majority of Africans would take a safe and effective vaccine. Nevertheless, vaccine hesitancy towards COVID-19 vaccines evolves over-time. In this view, it is crucial to investigate in depth barriers and facilitators influencing vaccine hesitancy/acceptability within African population.

During the last decade several initiatives have emerged that aim at improving vaccine coverage and acceptability across the African continent. A noteworthy example is the Francophone African Civil Society Organizations' Platform for Strengthening Health Systems and Immunization, which has been since 2015 supported by GAVI (Global Alliance for Vaccines and Immunisation). OAFRESS encourages activities among francophone African members, with the primary objective of reinforcing capacities and coordinating strategies among these countries. The last West African Ebola epidemic demonstrated the importance of engaging communities in order to promote vaccine acceptability. The three most hit countries, Guinea, Sierra Leone, and Liberia, worked together and invested in research and campaigns to identify and address barriers and facilitators of vaccine acceptance, which informed both clinical vaccine studies and roll-out strategies.

In order to promote the equitable and prompt roll-out of the COVID-19 vaccine worldwide, as the COVAX initiative strives for, factors influencing vaccine hesitancy in low and middle-income countries need to be investigated more thoroughly. The request for a first roll-out of the vaccines in eligible countries was to be submitted by December 7, 2020. Many of the eligible African countries have placed the order to receive the vaccines, which are already being deployed within these first months of 2021. Country and population preparedness are crucial to making the roll-out a success.

2. Study Objectives 2.1 Overall objective To investigate COVID-19 vaccine hesitancy among five African countries to inform effective context-specific public health strategies for roll-out of vaccination.

2.2 Primary objectives • To describe and compare levels of COVID-19 vaccine hesitancy among the general population and health care workers in rural and urban settings across African countries

2.3 Secondary objectives

• To explore factors influencing COVID-19 vaccination hesitancy among the general population and health care workers in urban and rural Africa

3. Methodology 3.1 Study design A cross-sectional survey will be conducted in five African countries. A core study will be implemented in five countries, other countries will enter the study as budget will become available. Study participants will be selected among the general population aged older than 18 and health care workers. Sample sizes have been calculated separately for these two groups.

ELIGIBILITY:
Inclusion Criteria:

General population

* Be at least 18 years of age, be willing and able to provide written informed consent AND

Health professionals

* To be health professionals working in health care institutions at all levels of care for the Ministry of Health (MoH)
* freely consent to participate in the study

Exclusion Criteria:

* All minors (<18)
* All individuals who do not meet the inclusion criteria listed above and those who are not willing to give written informed consent for participation in this research

In Senegal

* All those already vaccinated or being offered a vaccination for COVID-19 and refused and/or delayed the vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The general population will be selected in the capital and a rural area (around the capital) from each country. Approximately 5 clusters per area will be considered. The interviews will be house hold based.
  Health workers will be interviewed in facilities located in the study area and selected by the local study coordinator. Only people who have direct contact with patients will be considered for the analysis. To select study participants, staff lists including social workers from each facility will be used to randomly select people to be interviewed.
Sampling Method: Probability Sample
Enrollment: 4977 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine hesitancy | 1 month
  To describe and compare levels of COVID-19 vaccine hesitancy among the general population and health care workers in rural and urban settings across different African countries

SECONDARY OUTCOMES:
Factors influencing vaccine hesitancy | 1 month
  To explore factors influencing COVID-19 vaccination hesitancy among the general population and health care workers in urban and rural Africa

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Fusco, PhD, Principal Investigator — Bernhard Nocht Institute for Tropical Medicine; Henri Gautier Ouedraogo, Prof, Principal Investigator — University of Ouagadougu; Alpha Mahmoud Barry, Dr, Principal Investigator — Santé Plus; Seydou Doumbia, Prof, Principal Investigator — University of Bamako; Sylvain Faye, Prof, Principal Investigator — Cheikh Anta Diop University, Senegal; Abdullah Mbawah, Dr, Principal Investigator — University of Freetown
Locations (5):
- Henri Gautier Ouedragogo, Ouagadougou, Burkina Faso
- Alpha Mahmoud Barry, Conakry, Guinea
- Seydou Doumbia, Bamako, Mali
- Sylvain Faye, Dakar, Senegal
- Abdul Mbawah, Freetown, Sierra Leone

REFERENCES:
- [Background] MacDonald NE; SAGE Working Group on Vaccine Hesitancy. Vaccine hesitancy: Definition, scope and determinants. Vaccine. 2015 Aug 14;33(34):4161-4. doi: 10.1016/j.vaccine.2015.04.036. Epub 2015 Apr 17. PMID 25896383
- [Background] Lazarus JV, Ratzan SC, Palayew A, Gostin LO, Larson HJ, Rabin K, Kimball S, El-Mohandes A. A global survey of potential acceptance of a COVID-19 vaccine. Nat Med. 2021 Feb;27(2):225-228. doi: 10.1038/s41591-020-1124-9. Epub 2020 Oct 20. PMID 33082575
- [Background] Schwarzinger M, Watson V, Arwidson P, Alla F, Luchini S. COVID-19 vaccine hesitancy in a representative working-age population in France: a survey experiment based on vaccine characteristics. Lancet Public Health. 2021 Apr;6(4):e210-e221. doi: 10.1016/S2468-2667(21)00012-8. Epub 2021 Feb 6. PMID 33556325
- [Background] Samarasekera U. Feelings towards COVID-19 vaccination in Africa. Lancet Infect Dis. 2021 Mar;21(3):324. doi: 10.1016/S1473-3099(21)00082-7. No abstract available. PMID 33639125
- [Background] Dada S, McKay G, Mateus A, Lees S. Lessons learned from engaging communities for Ebola vaccine trials in Sierra Leone: reciprocity, relatability, relationships and respect (the four R's). BMC Public Health. 2019 Dec 11;19(1):1665. doi: 10.1186/s12889-019-7978-4. PMID 31829223
- [Background] Larson HJ, Jarrett C, Schulz WS, Chaudhuri M, Zhou Y, Dube E, Schuster M, MacDonald NE, Wilson R; SAGE Working Group on Vaccine Hesitancy. Measuring vaccine hesitancy: The development of a survey tool. Vaccine. 2015 Aug 14;33(34):4165-75. doi: 10.1016/j.vaccine.2015.04.037. Epub 2015 Apr 18. PMID 25896384
- [Derived] Di Meglio F, Lhomme E, Ouedraogo HG, Barry AM, Doumbia S, Faye SL, Mbawah AK, Sagna T, Tounkara M, Strauss R, Doumbia CO, Diouf S, Cisse K, May J, Puradiredja DI, Fusco D. Variations in COVID-19 vaccine hesitancy over time: a serial cross-sectional study in five West African countries. BMJ Open. 2024 Nov 7;14(11):e083766. doi: 10.1136/bmjopen-2023-083766. PMID 39510778
- [Derived] Faye SLB, Krumkamp R, Doumbia S, Tounkara M, Strauss R, Ouedraogo HG, Sagna T, Barry AM, Mbawah AK, Doumbia CO, Diouf S, Cisse K, Harding M, Donven P, May J, Puradiredja DI, Fusco D; ACHES consortium. Factors influencing hesitancy towards adult and child COVID-19 vaccines in rural and urban West Africa: a cross-sectional study. BMJ Open. 2022 Apr 13;12(4):e059138. doi: 10.1136/bmjopen-2021-059138. PMID 35418436